CLINICAL TRIAL: NCT00599872
Title: Parallel, Randomized, Double-Blind, Placebo-Controlled Trial in Adults for the Sublingual-Oral Immunotherapy (SLIT) of Allergic Rhinoconjunctivitis With or Without Asthma Caused By Ragweed Pollen
Brief Title: Efficacy Study of Sublingual Immunotherapy to Treat Ragweed Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Greer Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLIT07-01
Record Dates: First submitted 2007-12-20; First posted 2008-01-24 (Estimated); Results first posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2014-12

CONDITIONS: Allergic Rhinitis
Keywords: Allergy; Sublingual Immunotherapy; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ragweed Allergenic Extract (Active Comparator): Standardized Ragweed Allergenic Extract administered via the sublingual oral route (27.6 to 77.3 Amb a 1 Units)
  Interventions: Biological: Standardized Ragweed Allergenic Extract
- Placebo (Placebo Comparator): Standardized Ragweed Allergenic Extract Placebo via the sublingual oral route
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Standardized Ragweed Allergenic Extract — Standardized Ragweed Allergenic Extract, sublingual oral
  Arms: Ragweed Allergenic Extract
Biological: Placebo — Placebo, sublingual oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine an effective dose range for the administration of ragweed allergenic extract via the sublingual route of administration

DETAILED DESCRIPTION:
Specific allergen immunotherapy as currently practiced in the USA and described in product labeling comprises the subcutaneous injection of incrementally increasing doses to a targeted maintenance dose ("build-up") followed by maintenance injections of allergenic extract/vaccine. Up to 30-40 injections may be required during the build-up phase over a 3-6 month period. When adequate maintenance doses are reached, this form of immunotherapy (SCIT) has been shown to be highly effective and safe.

Standard practices recommend that the injections be given under the supervision of trained physicians and that the patient remain in the physician's office at least 20 to 30 minutes after an injection. The administration of immunotherapy injections are not recommended at home because of the risk of inadequate recognition and treatment of systemic reactions. The inconvenience and expense of traveling for allergy injections and the discomfort of the repeated injections is a disincentive to this form of treatment particularly in pediatric patients. For example, dropout rates exceeding 50% over a multi-year course of injection treatment have been reported.

Alternative routes for immunotherapy have been explored, especially in Europe in an attempt to improve patient compliance and to minimize the risk of serious adverse reactions. For example, sublingual-oral immunotherapy (SLIT), which is the administration of the allergenic extract/vaccine under the tongue for 1-2 minutes followed by swallowing, has been proven to be efficacious and safe in several double-blind, placebo-controlled studies. A recent Cochrane Review concluded, "SLIT is a safe treatment, which significantly reduces symptoms and medication requirements in allergic rhinitis."

Efficacy studies support the use of SLIT for the treatment of rhinitis or rhinitis and asthma. However, dosage schedules are highly variable and optimal maintenance doses have not yet been established. Thus, dosing studies should be designed to investigate not only the safety profile but to determine optimal doses for maintenance therapy of patients built-up by injection IT and for build-up regimens of previously untreated patients.

Much of the United States medical community's hesitation to embrace sublingual immunotherapy as a viable treatment option for allergy patients has stemmed from limited information using U.S. licensed allergenic extracts for this treatment route. Additionally, the cost-effectiveness of one form of therapy over the other has not been clearly evaluated and the third-party payers have not accepted SLIT for insurance coverage.

ELIGIBILITY:
Inclusion Criteria:

* Adult ragweed-sensitive Subjects with allergic rhinoconjunctivitis with or without asthma during ragweed pollen season.
* Subjects must be 18 to 50 years of age.
* Test Subjects will have a history of moderate to severe isolated or unseasonal allergic rhinoconjunctivitis with or without mild intermittent asthma symptoms attributable to ragweed pollen for a minimum of 2 years before study entry.
* Subjects with or with out a history of asthma will possess FEV1 and PEF greater than or equal to 80% predicted at the beginning of the study established by spirometry and defined by the Knudson predicted set.
* Sensitivity to the relevant allergen will be documented by a positive skin prick test result performed along with negative (saline) and positive (histamine) control skin tests. A positive test will be defined as the skin reaction having the longest wheal diameter of 5mm or greater or the longest erythema diameter of 10 mm or greater at 15-20 minutes after application.
* All female Subjects of child-bearing potential will be required to provide a urine sample for pregnancy testing that must be negative before being allowed to participate in the study.
* Subjects must be planning to remain in the study area during the trial (see exclusion criteria # 14).
* Subjects must be trained on the proper use of the EpiPen, and sign the EpiPenTraining Form before being allowed to enroll in the study.
* Subjects must be mentally and physically capable of self-administering oral drug.

Exclusion Criteria:

* Subjects having a history of anaphylaxis or history consistent with persistent asthma
* Subjects taking antihistamines or nasal steroids medications greater than twice a week in the months of January and/or February.
* Subjects with chronic sinusitis unstable angina, significant arrhythmia, uncontrolled hypertension, or other chronic or immunological diseases that in the opinion of the investigator might interfere with the evaluation of the test drug or pose additional risk to the Subject.
* Subjects having perennial or structurally related rhinitis or rhinitis medicamentosa (from excessive use of nasal decongestants) that will interfere with the evaluation of symptoms due to ragweed allergy.
* Subjects with an FEV1 or PEF less than 80% predicted (moderate persistent asthma) with or without controller medication.
* Subjects who have received an experimental drug in the 30 days prior to admission into this study or who plan to use an experimental drug during the study.
* Subjects who have received Anti-IgE medications (Xolair) or similar compounds in the last 12 months.
* Subjects who have received ragweed allergen immunotherapy in the last 3 years prior to admission into this study.
* Subjects who are current users of inhaled, oral, intramuscular, intravenous corticosteroids, tricyclic antidepressants, beta blockers, or MAO inhibitors.
* Subjects using beta-agonist more than twice a month unless being taken prior to exercise.
* Subjects using medications that could induce adverse gastrointestinal reactions during the study. Subjects using such medications must prove stable with no side effects for at least 3 months prior to enrollment.
* Subjects refusing to sign the EpiPen Training Form will be excluded from the study.
* Pregnant or breast feeding females.
* Subjects who plan to leave the study area for more than 2 consecutive weeks during the study.
* Subjects with a positive skin prick test to cat and/or dog, and own the pet(s) to which they are allergic.
* Subjects who sleep during the day due to working third shift.
* Subjects unable to achieve dose #2 or higher during preliminary dosing will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 430 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Esch, PhD, Study Director — Greer Laboratories, Inc.
Locations (30):
- United States (30):
  - Sneeze, Wheeze, & Itch Associates, Normal, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Iowa Clinical Research Corporation, Iowa City, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - College Park Family Care Center, Overland Park, Kansas
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - Family Allergy and Asthma Respiratory Institute, Louisville, Kentucky
  - Clinical Research Institute, Minneapolis, Minnesota
  - Clinical Research of the Ozarks, Rolla, Missouri
  - Midwest Clinical Research, LLC, St Louis, Missouri
  - Asthma, Immunology and Allergy Association, LLC, Lincoln, Nebraska
  - Midwest Allergy and Asthma Clinic, PA, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska
  - Ocean Allergy and Respiratory Research Center, Brick, New Jersey
  - Pulmonary and Allergy Associates, PA, Summit, New Jersey
  - Allergy and Respiratory Center, Canton, Ohio
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Oklahoma Allergy & Asthma Clinic, PC, Oklahoma City, Oklahoma
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - Allergy and Asthma Specialists, PC, Blue Bell, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - Vanderbilt ASAP Research, Nashville, Tennessee
  - Pharmaceutical Research & Consulting, Inc, Dallas, Texas
  - Allergy, Asthma and Sinus Center, SC, Greenfield, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
  - Aurora Advanced Healthcare, Inc, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Ragweed allergenic extract administer once daily at 77.3 Units/Amb a 1.
- Placebo: Placebo to be administered once daily at 0.0 Units/Amb a 1
Period: Overall Study
Arm/Group | Active | Placebo
Started | 216 | 214
Completed | 167 | 181
Not Completed | 49 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Placebo | Total
Number analyzed (Participants) | 216 | 214 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 216 | 214 | 430
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (9.54) | 35.5 (9.24) | 35.6 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 127 | 265
  Male | 78 | 87 | 165
Region of Enrollment [Number; unit: participants]
  United States | 216 | 214 | 430

OUTCOME MEASURES:

1. Primary Outcome: Scores on a Scale (Average of Daily Rhinoconjunctivitis Symptom Score (RSS) Recorded During the Ragweed Season
Description: Symptom score defined as sum of scores from eight symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe): ocular (itchiness, swelling/redness, and watery eyes/tears), nasal (sneezing, itching, runny and stuffy nose), and ears (itching). Average daily RSS ranged from 0-48; A lower score was more favorable.
  The average daily RSS was computed for each subject by: (1) summing the 8 individual allergy symptoms recorded in the morning (AM RSS) and the evening (PM RSS); (2) forming the daily RSS by summing the AM RSS and the PM RSS for each day of the ragweed season; (3) averaging the daily RSS for the entire ragweed pollen season.
Time Frame: Ragweed pollen season, 08/01/08 to 10/30/08, approximately 3 months
Population: The modified ITT population: subjects with 12 weeks or more of treatment (based on subject consent date and date of ragweed season for the site)
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Active: Ragweed allergenic extract administer once daily at 26.3 to 77.3 Units/Amb a 1.
Arm/Group | Active | Placebo
Number analyzed (Participants) | 136 | 157
Scores on a scale | 6.2 (6.2) | 6.5 (5.61)
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = -0.418, 95% CI 2-sided [-1.15 to 0.48]

2. Secondary Outcome: Scores on a Scale (Average Daily RSS During the Highest Pollen Count Week)
Description: Symptom score defined as sum of scores from eight symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe): ocular (itchiness, swelling/redness, and watery eyes/tears), nasal (sneezing, itching, runny and stuffy nose), and ears (itching). Average daily RSS ranged from 0-48; A lower score was more favorable.
  The average daily RSS was computed for each subject by: (1) summing the 8 individual allergy symptoms recorded in the morning (AM RSS) and the evening (PM RSS); (2) forming the daily RSS by summing the AM RSS and the PM RSS for each day of the ragweed season; (3) averaging the daily RSS for the entire ragweed pollen season.
  The highest pollen count week was defined as the 7 contiguous days from the series with the largest average pollen count, and in which the weekly average was computed using at least 4 non-missing daily RSS values (either AM or PM could be present to be considered a valid daily RSS value).
Time Frame: 09/01/2008-09/07/2008
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: scores on a scale
Groups:
- Active: Ragweed allergenic extract administer once daily at 27.6 to 77.3 Units/Amb a 1.
Arm/Group | Active | Placebo
Number analyzed (Participants) | 136 | 157
scores on a scale | 7.0 (6.96) | 7.5 (7.03)
Statistical Analysis 1: Comparison: Active vs Placebo; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Net) = 0.360, 95% CI 2-sided [-1.72 to 0.63]

3. Secondary Outcome: Scores on a Scale (Average Daily AM RSS and the Average Daily PM RSS During the Ragweed Season)
Description: Symptom score defined as sum of scores from eight symptoms rated 0-3 (0=absent, 1=mild, 2=moderate, 3=severe): ocular (itchiness, swelling/redness, and watery eyes/tears), nasal (sneezing, itching, runny and stuffy nose), and ears (itching). Average daily RSS ranged from 0-48; A lower score was more favorable.
  The average daily RSS (the sum of the 8 individual allergy symptoms recorded in the morning (AM RSS) and the evening (PM RSS).
Time Frame: Ragweed pollen season 08/01/08 to 10/30/08
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ragweed Allergenic Extract | Placebo
Number analyzed (Participants) | 136 | 157
Scores on a scale
  Average Daily AM RSS | 3.5 (3.64) | 3.8 (3.22)
  Average Daily PM RSS | 3.5 (3.47) | 3.6 (3.11)

4. Secondary Outcome: Scores on a Scale (Average Daily RSS During the Ragweed Season for Each of the Three Organ) Systems (Ocular, Nasal, Ears);
Description: The average daily RSS during the ragweed season for each of the 3 organ systems (ocular, nasal, ears) were separately analyzed to evaluate these individual components of the RSS. Three separate baseline average daily RSS values were computed for this analysis. The modified ITT population was used for this analysis. The range for scores: 0 to 3 for each of eight symptom or a total of 0 to 24 daily RSS. A lower score was more favorable.
Time Frame: Ragweed pollen season 08/01/08 to 10/30/08
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 136 | 157
Scores on a scale
  Ocular | 1.7 (2.44) | 1.9 (2.12)
  Nasal | 4.0 (3.55) | 4.2 (3.41)
  Ears | 0.5 (0.94) | 0.5 (0.70)

5. Secondary Outcome: Scores on a Scale (Total Allergy Relief Medication Score During the Ragweed Season) for Each Subject
Description: Total allergy relief medication score during the ragweed season for each subject. This score is computed for each subject by summing their individual medication scores (excluding beta-agonist use) for the entire ragweed season. High scores were indicative of poor symptom relief from the study medication. The associated relief medication scores assigned to medication are 0-if no medication taken; 3 for each one antihistamine tablet taken; 1 for each 2 antihistamine eye drop administrations, 1 for each 2 antihistamine nasal spray administrations and 1 for each puff of beta-agonist. The maximum medication score was dependent on the cumulative rescue medication use. The lower result the more favorable.
Time Frame: Ragweed pollen season 08/01/08 to 10/30/08
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 136 | 157
Scores on a scale | 40.5 (85.59) | 50.1 (137.00)

6. Secondary Outcome: Scores on a Scale (The Average Combined Allergy Symptom and Medication Score During the Ragweed Season for Each Subject)
Description: The average combined allergy symptom and medication score during the ragweed season for each subject. This score is computed for each subject by adding their daily relief medication scores (excluding beta-agonist use) and their daily RSS for the entire ragweed season, and then taking the average of the combined scores across days.
Time Frame: Ragweed pollen season 08/01/08 to 10/30/08
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Active | Placebo
Number analyzed (Participants) | 136 | 157
Scores on a scale | 6.7 (6.85) | 7.3 (6.69)

ADVERSE EVENTS:
Time Frame: Approximately 30 weeks
Groups:
- Ragweed Allergenic Extract: Ragweed Allergenic extract administered once daily at 77.3 Units/Amb a 1.
- Placebo: Placebo be administered once daily at 0.0 Units/Amb a 1
Arm/Group | Ragweed Allergenic Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 3/216 | 0/214
Other Adverse Events (participants affected / at risk) | 0/216 | 0/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ragweed Allergenic Extract (N=216) | Placebo (N=214)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Stress (Psychiatric disorders) | 1 (1) | 0
food poisoning (Gastrointestinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No